CLINICAL TRIAL: NCT03646968
Title: Phase II Study to Evaluate the Effectiveness and Safety of Anlotinib Combined With Docetaxel in Progress After First Line Standard Cheomotherapy in Advanced Non-driver Mutation Non- Squamous Non-small Cell Lung Cancer
Brief Title: Study of Anlotinib Combined With Docetaxel in Non-Driver Mutation Non-squamous NSCLC: the Save Study
Acronym: SAVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yongchang Zhang (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAVE
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-Squamous Non Small Cell Lung Cancer
Keywords: Anlotinib Combined With Docetaxel
MeSH Terms: interventions — anlotinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohorts (Experimental): Phase II Study to evaluate the Effectiveness and Safety of Anlotinib combined with Docetaxel in Progress after First line Standard Cheomotherapy in advanced non-driver mutation non- squamous non-small cell lung cancer
  Interventions: Drug: Anlotinib and Docetaxel

INTERVENTIONS:
Drug: Anlotinib and Docetaxel — Patients who was Progress after First line Standard Cheomotherapy in advanced non-driver mutation non- squamous non-small cell lung cancer recieved the treatment of Anlotinib and Docetaxel (Anlotinib, 12mg, po,qd and Docetaxel 175mg/m2, ivgtt, every 21day)

SUMMARY:
The purpose of this study is to evaluate the Effectiveness and Safety of Anlotinib combined with Docetaxel in Progress after First line Standard Cheomotherapy in advanced non-driver mutation non- squamous non-small cell lung cancer

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Effectiveness and Safety of Anlotinib combined with Docetaxel in Progress after First line Standard Cheomotherapy in advanced non-driver mutation non- squamous non-small cell lung cancer .According to the result of TAX317,the ORR of second line standard chemotherapy was 5- 8%. We expect the ORR was 20%. Using PASS11, we calculated the sample size of this study was 39 , according to 10% censoring,the expected sample size is 43.

ELIGIBILITY:
Inclusion Criteria:

* 18，Pathologically proven Non squamous non small cell lung cancer

  * No-drive gene mutaion (EGFR、ALK、ROS1） by NGS
  * Progress after second line
  * PS score 0-2

Exclusion Criteria:

* Patients received second line treatment
* Patients received treatment of Anlotinib or Docetaxel
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | may 2018- may 2019 (1 year)
  overall response rate

SECONDARY OUTCOMES:
PFS | may 2018- may 2019 (1 year)
  Progression survival time
OS | may 2018- may 2019 (1 year)
  overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China